CLINICAL TRIAL: NCT05792995
Title: Foundation and Clinical About the Expression of PD-1 in Peripheral Blood T Lymphocytes and Its Prediction of Immune Efficacy of Patients With Non-small Cell Lung Cancer
Brief Title: Foundation and Clinical About the Expression of PD-1 in Peripheral Blood T Lymphocytes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Xin-Hua Xu (Other)
Responsible Party: Sponsor-Investigator, Xin-Hua Xu, professor, China Three Gorges University, Yichang, China
Organization: China Three Gorges University, Yichang, China (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CTGU007
Record Dates: First submitted 2023-03-11; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Nivolumab; durvalumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Immunomonotherapy plus Chemotherapy plus Anti-angiogenesis Therapy (Experimental): Any first-line treatment that includes immunotherapy.
  Interventions: Drug: Sindillimab
- Chemotherapy plus Immunomonotherapy (Experimental): Any first-line treatment that includes immunotherapy.
  Interventions: Drug: Sindillimab
- Immunomonotherapy plus Anti-angiogenesis Therapy (Experimental): Any first-line treatment that includes immunotherapy.
  Interventions: Drug: Sindillimab
- Immunomonotherapy (Experimental): Any first-line treatment that includes immunotherapy.
  Interventions: Drug: Sindillimab

INTERVENTIONS:
Drug: Sindillimab — Any treatment regimen that includes immunotherapy.
  Other Names: Pembrolizumab; Nivolumab; Durvalumab

SUMMARY:
Providing more theoretical basis for the prediction of the efficacy of advanced NSCLC and helping select better advantaged population of NSCLC immunotherapy to maximize the benefits of patients By exploring the relationship between the changes of PD-1 expression in peripheral blood T lymphocytes and the clinical efficacy before and after the use of PD-1 / PD-L1 inhibitors.

DETAILED DESCRIPTION:
From the perspective of immunology, it is intended to explore whether the expression of PD-1 in peripheral blood T lymphocytes can be used as a reference index for selecting immune "+" therapy in patients with advanced HCC, and to clarify the relationship between the expression level of peripheral blood T lymphocytes and the survival data of patients receiving immune "+" therapy. And explore whether there is consistency between the expression level of PD-L1 and that of PD-L1 on patients. At the same time, to explore whether there is a correlation between the distribution of T cell subsets and the efficacy of immunotherapy, so as to provide a new theoretical basis for the clinical screening of the target population of immune "+" therapy and a new clinical screening index for the prognosis assessment of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in clinical research; fully understand and know the research and sign informed consent.
2. Age ≥18 years, and ≤75years , either sex.
3. Eastern Collaborative Oncology Group Performance status (ECOG PS) 0 ,1 or 2.
4. Patients with NSCLC diagnosed by histopathology (according to the 8th edition of AJCC).
5. Initial diagnosis patients unable to perform surgery.
6. Normal hepatic function: total bilirubin≤1.5×normal upper limit (ULN); Alanine aminotransferase and Aspartate aminotransferase levels ≤2.5×ULN or ≤5×ULN if liver metastasis is present.
7. Normal renal function ：Creatinine ≤1.5×ULN or calculated creatinine clearance ≥45 mL/min (using Cockcroft/Gault formula to calculate ).
8. Normal hematological function：absolute neutrophil count ≥1.5×109/L, platelet count ≥70×109/L, hemoglobin≥80g/L [no blood transfusion or erythropoietin (EPO) within 7 days] Dependency].
9. Has a life expectancy of at ≥3 months.
10. EGFR and ALK were negative.

Exclusion Criteria:

1. ECOG PS >2.
2. Patients who received radiotherapy, chemotherapy, monoclonal antibody and oral EGFR-TKI therapy within six months.
3. Patients who are receiving any other investigational agents within 30 days prior to entering the study.
4. History of other malignancies (except for cured cervical carcinoma in situ or skin basal cell carcinoma and other malignancies that have been cured for more than 5 years).
5. Have no measurable lesion as defined by RECIST 1.1.
6. Accompanied by other serious diseases, including but not limited to:

   Uncontrollable congestive heart failure (NYHA grade Ⅲ or Ⅳ), unstable angina, poorly controlled arrhythmia, uncontrolled moderate or above hypertension (SBP > 160mmhg or DBP > 100mmhg) ; Severe active infection; Uncontrollable diabetes (refers to the high fluctuation of blood glucose, the impact on patients' life and the frequent occurrence of hypotension despite the standard insulin treatment and frequent blood glucose monitoring) ; Mental illness affecting informed consent and / or program compliance.
7. Those who are allergic to the drug or its components used in the program.
8. Pregnancy (confirmed by hCG test in blood or urine) or lactating women, or childbearing age subjects are unwilling or unable to take effective contraceptive measures (applicable to both male and female subjects) until at least 6 months after the last trial treatment.
9. Those who are not considered suitable for the study by the researchers.
10. Unwilling to participate in this study or unable to sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Compare Progression Free Survival (PFS) Regimen using RECIST 1.1. | approximately 24 months
  PFS was defined as the time between the date of randomization and the date of first documented disease progression or death, whichever occurs first. Disease progression was determined based on investigator assessment using response evaluation criteria In solid tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Compare Overall Survival (OS) | approximately 24 months
  Overall Survival (OS) was defined as the time from the date of randomization to the date of death due to any cause. Data for participants who were not reported as dead at the time of analysis was censored at the date when they were last known to be alive.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Central Hospital of Yichang City, the First Clinical Medical College of Three Gorges University, Yichang, Hubei, China